CLINICAL TRIAL: NCT05938725
Title: KYSA-1: A Phase 1/2, Open-Label, Multicenter Study of KYV-101, an Autologous Fully-Human Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Refractory Lupus Nephritis
Brief Title: KYSA-1: A Study of Anti-CD19 Chimeric Antigen Receptor T-Cell (CD19 CAR T) Therapy, in Subjects With Refractory Lupus Nephritis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kyverna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KYSA-1; KYV101-001 (Other: Kyverna Therapeutics)
Record Dates: First submitted 2022-10-11; First posted 2023-07-10 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Lupus Nephritis; Lupus Nephritis - World Health Organization (WHO) Class III; Lupus Nephritis - WHO Class IV
Keywords: KYV-101; glomerulonephritis; autoimmune disease; anti-CD19 CAR-T therapy; cellular therapy
MeSH Terms: conditions — Lupus Nephritis; Glomerulonephritis; Autoimmune Diseases | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- KYV-101 CAR-T cells with lymphodepletion conditioning (Phase 1) (Experimental): Dosing with KYV-101 CAR T cells
  Interventions: Biological: KYV-101 anti-CD19 CAR-T cell therapy; Drug: Standard lymphodepletion regimen
- KYV-101 CAR-T cells with lymphodepletion conditioning (Phase 2) (Experimental): Recommended Phase 2 Dose
  Interventions: Biological: KYV-101 anti-CD19 CAR-T cell therapy; Drug: Standard lymphodepletion regimen

INTERVENTIONS:
Biological: KYV-101 anti-CD19 CAR-T cell therapy — KYV-101 anti-CD19 CAR-T cell therapy
Drug: Standard lymphodepletion regimen — Standard lymphodepletion regimen
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
A Study of Anti-CD19 Chimeric Antigen Receptor T Cell Therapy for Subjects With Refractory Lupus Nephritis

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease characterized by a wide spectrum of organ involvement and disease severity. Renal involvement (categorized as lupus nephritis [LN]) may occur in approximately 50% of SLE patients and is marked by proteinuria, microscopic hematuria, and varying degrees of renal insufficiency. B cells play a central role in the pathogenesis of SLE and LN, with autoantibodies developing as an early finding, and local, tissue resident B cells producing pathogenic autoantibodies and driving inflammation and tissue damage over time. CD19-targeted chimeric antigen receptor (CAR) T cells harness the ability of cytotoxic T cells to directly and specifically lyse target cells to effectively deplete B cells in the circulation and in lymphoid and potentially non-lymphoid tissues. KYV-101, a fully human anti-CD19 CAR T-cell therapy, will be investigated in adult subjects with refractory lupus nephritis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Clinical diagnosis of SLE according to 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) classification criteria
3. Biopsy-proven proliferative LN Class III or IV according to 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria
4. Positive anti-nuclear antibody (ANA) (titer ≥1:80 ), anti-dsDNA (≥30 IU/mL on enzyme-linked immunosorbent assay [ELISA]), or anti-Smith at screening or by documented medical history
5. Up to date on recommended vaccinations, including against coronavirus disease 2019 (COVID-19)/ severe acute respiratory syndrome coronavirus 2 (SARS-Cov-2), per Centers for Disease Control and Prevention (CDC) or institutional guidelines for immune compromised individuals

Exclusion Criteria:

1. Rapidly progressive glomerulonephritis; history of or currently active severe central nervous system (CNS) lupus, including cerebritis, cerebrovascular accident, and seizures
2. Prior treatment with cellular immunotherapy (CAR-T) or gene therapy product directed at any target
3. History of allogeneic or autologous stem cell transplant
4. Evidence of active hepatitis B or hepatitis C infection
5. Positive serology for HIV
6. Primary immunodeficiency
7. History of splenectomy
8. History of stroke, seizure, dementia, Parkinson's disease, coordination movement disorder, cerebellar diseases, psychosis, paresis, aphasia, and any other neurologic disorder investigator considers would increase the risk for the subject
9. Impaired cardiac function or clinically significant cardiac disease
10. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to screening)
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to screening
    3. A primary malignancy which has been completely resected, or treated, and is in complete remission for at least 5 years prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence adverse events (AEs) and laboratory abnormalities (Phase 1 and Phase 2) | Up to 2 years
Frequency of dose limiting toxicities at each dose level (Phase 1) | Up to 2 years
To Evaluate efficacy (Phase 2) | Up to 52 Weeks
  Complete renal response rates (CRR)

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) (Phase 1 and Phase 2) | Up to 2 years
  Levels of KYV-101 CAR-positive T cells in the blood
To characterize the pharmacodynamics (PD) (Phase 1 and Phase 2) | Up to 2 years
  Levels of B cells in the blood
To characterize the pharmacodynamics (PD) (Phase 1 and Phase 2) | Up to 2 months
  Levels of cytokines in serum
To evaluate disease related biomarkers (Phase 1 and Phase 2) | Up to 2 years
  Levels of anti-double stranded DNA (anti-dsDNA) in serum
To evaluate disease related biomarkers (Phase 1 and Phase 2) | Up to 2 years
  Levels of complement C3, C4 in serum
To evaluate efficacy (Phase 1 and Phase 2) | 12, 24, and 52 weeks
  Complete renal response rates (CRR)
To evaluate efficacy (Phase 1 and Phase 2) | Up to 2 years
  Time to Complete renal response rates (CRR)
To evaluate efficacy (Phase 1 and Phase 2) | Up to 2 years
  Time from first achieved CRR to disease worsening or end of study
To evaluate efficacy (Phase 2) | Up to 52 weeks
  Duration of CRR to Week 52 but no less than 12 weeks (duration of remission)
To evaluate the immunogenicity (humoral response) of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Percentage of participants who develop anti-KYV-101 antibodies by immunoassays
To assess PRO after infusion of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Change from Baseline in SF-36
To assess PRO after infusion of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Change from Baseline in FACIT-F
To assess PRO after infusion of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Change from Baseline in Lupus QoL Questionnaire
To assess PRO after infusion of KYV-101 (Phase 1 and Phase 2) | Up to 2 years
  Change from Baseline in WPAI
To define the Recommended Phase 2 Dose (RP2D) (Phase 1) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Kyverna Therapeutics
Locations (6):
- United States (6):
  - Stanford University Medical Center, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - University of Massachusetts Worcester, Worcester, Massachusetts
  - Northwell Health, Great Neck, New York
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brudno JN, Lam N, Vanasse D, Shen YW, Rose JJ, Rossi J, Xue A, Bot A, Scholler N, Mikkilineni L, Roschewski M, Dean R, Cachau R, Youkharibache P, Patel R, Hansen B, Stroncek DF, Rosenberg SA, Gress RE, Kochenderfer JN. Safety and feasibility of anti-CD19 CAR T cells with fully human binding domains in patients with B-cell lymphoma. Nat Med. 2020 Feb;26(2):270-280. doi: 10.1038/s41591-019-0737-3. Epub 2020 Jan 20. PMID 31959992
- [Background] Mackensen A, Muller F, Mougiakakos D, Boltz S, Wilhelm A, Aigner M, Volkl S, Simon D, Kleyer A, Munoz L, Kretschmann S, Kharboutli S, Gary R, Reimann H, Rosler W, Uderhardt S, Bang H, Herrmann M, Ekici AB, Buettner C, Habenicht KM, Winkler TH, Kronke G, Schett G. Anti-CD19 CAR T cell therapy for refractory systemic lupus erythematosus. Nat Med. 2022 Oct;28(10):2124-2132. doi: 10.1038/s41591-022-02017-5. Epub 2022 Sep 15. PMID 36109639